CLINICAL TRIAL: NCT01021397
Title: Phase I Study to Determine the Safety, Infectivity, and Tolerability of 2 Doses of Live Attenuated Recombinant Cold-Passaged (cp) 45 Human Parainfluenza Type 3 Virus Vaccine, rHPIV3cp45, Lot PIV3#102A, Delivered as Nose Drops to HPIV3-Seronegative Infants and Children 6 to 36 Months of Age, at a 6 Month Interval
Brief Title: Safety of and Immune Response to Recombinant Live Attenuated Parainfluenza Type 3 Virus Vaccine in Healthy Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 255
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Paramyxoviridae Infections; Virus Diseases
Keywords: Respiratory Tract Infection
MeSH Terms: conditions — Paramyxoviridae Infections; Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive one dose of vaccine virus at study entry and between Weeks 22 and 27
  Interventions: Drug: rHPIV3cp45
- 2 (Placebo Comparator): Participants will receive one dose of vaccine virus placebo at study entry and between Weeks 22 and 27
  Interventions: Drug: rHPIV3cp45 placebo

INTERVENTIONS:
Drug: rHPIV3cp45 — 10^5 TCID50 nasal drops
  Arms: 1
Drug: rHPIV3cp45 placebo — 1X-L15 nasal drops
  Arms: 2

SUMMARY:
Human parainfluenza viruses (HPIVs) are a major health concern in infants and young children under 5 years of age, causing serious respiratory tract disease. The primary purpose of this study is to test the safety of and immune response to a new HPIV vaccine in healthy infants and children.

DETAILED DESCRIPTION:
HPIV type 3 (HPIV3) ranks second only to respiratory syncytial virus as the most important cause of bronchiolitis and pneumonia in infants less than 6 months of age. HPIV3 can cause severe disease in the first 2 years of life and is responsible for 11% of hospitalizations for respiratory diseases in children. This study will evaluate the safety and immunogenicity of a live recombinant attenuated intranasal HPIV3 vaccine, rHPIV3cp45.

This study will last for approximately 28 weeks. Infants and children 6 months to 36 months of age will be randomly assigned to one of two groups. Group 1 participants will receive 2 immunizations of rHPIV3cp45. Group 2 participants will receive 2 doses of rHPIV3cp45 placebo. Immunizations will be given as nose drops and administered at study entry and approximately 22 to 27 weeks after study entry.

On the day of immunization, a physical exam and blood collection will occur. Participants will be observed for 15 minutes after immunization for any immediate adverse effects. Parents or guardians will be given a thermometer to take with them and will be instructed on how to take their child's temperature. They will be given the study schedule and will need to provide contact phone numbers so study personnel can contact them by phone during the days after immunization. Parents and guardians will be contacted by telephone daily from Day 1 to Day 18 after each immunization.

Parents or guardians will need to record their child's temperature daily for at least 17 days immediately following immunization. During this 17-day period, study visits will occur on Days 3, 6, and 12 after each dose of vaccine or placebo. Participants will undergo a nasal wash for a viral culture at all study visits. There will be additional follow-up visits occurring sometime between 49 and 63 days after the first dose and 28 to 35 days after the second dose; blood collection will occur at the follow-up visits. Additional visits may be required on selected days during the month after immunization. Infants who experience illness or side effects may be asked to return to the clinic for examination.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* HPIV3-uninfected
* Has received age-appropriate inactivated or subunit routine immunizations at least 2 weeks prior to study entry
* Has received age-appropriate live routine immunizations at least 4 weeks prior to study entry and at least 2 weeks for rotavirus and inactivated vaccines
* Available for the duration of the trial
* Parent or guardian reachable by telephone for post-immunization contact
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Known or suspected impairment of immunologic functions. Infants who are HIV-infected, who are bone marrow or solid organ transplant recipients, or who have received immunosuppressive therapy, including systemic corticosteroids within 30 days prior to study entry. Infants who are using topical steroids, topical antibiotic ointments and topical antifungal agents are not excluded.
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previously received HPIV3 vaccine
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including reactive airway disease. Infants with clinically insignificant cardiac abnormalities are not excluded. Infants or children who wheezed once or received bronchodilator therapy once in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months are not excluded.
* Born prematurely before the 37th week of pregnancy if participant is currently less than 12 months of age
* Member of a household containing immunocompromised individuals, pregnant caregivers, or infants less than 6 months of age
* Attends day care with infants less than 6 months of age
* Parent or guardian unable or unwilling to suspend daycare for 14 days following each immunization. More information on this criterion can be found in the protocol.
* Enrolled in another investigational drug or vaccine study from 30 days prior to study entry until the final follow-up blood draw

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events and other adverse events | Throughout study
Amount of serum antibody induced by vaccine in each recipient | Throughout study

SECONDARY OUTCOMES:
Amount of vaccine virus shed by each recipient | Throughout study
Immunogenicity of a second dose of vaccine and the protection of the first dose against re-infection with the second dose | From Weeks 22 to 28
Number of vaccinated infants infected with rHPIV3cp45 | Throughout study
Number of vaccinated participants infected with a second dose of rHPIV3cp45 | From Weeks 22 to 28
Phenotypic stability of vaccine virus shed | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Study Chair — Center for Immunization Research, Johns Hopkins University School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR), Johns Hopkins School of Public Health, Baltimore, Maryland
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Madhi SA, Cutland C, Zhu Y, Hackell JG, Newman F, Blackburn N, Murphy BR, Belshe RB, Karron RA, Deatly AM, Gruber WC, Bernstein DI, Wright PF. Transmissibility, infectivity and immunogenicity of a live human parainfluenza type 3 virus vaccine (HPIV3cp45) among susceptible infants and toddlers. Vaccine. 2006 Mar 20;24(13):2432-9. doi: 10.1016/j.vaccine.2005.12.002. Epub 2005 Dec 20. PMID 16406170
- [Background] Skiadopoulos MH, Surman SR, Riggs JM, Orvell C, Collins PL, Murphy BR. Evaluation of the replication and immunogenicity of recombinant human parainfluenza virus type 3 vectors expressing up to three foreign glycoproteins. Virology. 2002 May 25;297(1):136-52. doi: 10.1006/viro.2002.1415. PMID 12083844